CLINICAL TRIAL: NCT02096679
Title: A Phase I, Single-centre, Non-Randomised, Open-label, Pharmacokinetic and Mass Balance Study of Orally Administered [14C]-AZD9291 in Healthy Male Volunteers
Brief Title: Study Evaluating the Pharmacokinetic and Mass Balance of Single Dose [14C] AZD9291 in Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D5160C00011
Record Dates: First submitted 2014-03-24; First posted 2014-03-26 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Healthy Volunteers
Keywords: Phase I, healthy, pharmacokinetics, Mass balance
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-AZD9291 20mg (oral solution) (Experimental): Volunteers will receive 20 mg [14C]-AZD9291 containing a nominal 1 μCi activity, administered by mouth, as a solution.
  Interventions: Drug: AZD9291

INTERVENTIONS:
Drug: AZD9291 — Volunteer will receive a single oral dose of 20 mg [14C]-AZD9291 as a solution on Day 1

SUMMARY:
Study to evaluate the pharmacokinetic and Mass Balance of single dose [14C] AZD9291 in healthy male volunteers

DETAILED DESCRIPTION:
A Single-centre, Non-Randomised, Open-label, Pharmacokinetic and Mass Balance Study of Orally Administered [14C]-AZD9291 in Healthy Male Volunteers

ELIGIBILITY:
Inclusion Criteria:

1, Volunteers must be willing to use reliable methods of contraception (condom and spermicide), even if their partners are postmenopausal, surgically sterile, or using an effective hormonal method of contraception or intrauterine coil. 2. In addition, volunteers must agree to continue to take similar contraceptive precautions until 6 months after the last administration of AZD9291 and avoid procreative sex as well as sperm donation for 6 months.

Exclusion Criteria: 1, Any clinically relevant abnormalities in physical examination, vital signs, hematology,clinical chemistry, urinalysis or ECG at baseline in the opinion of the investigator. 2. Radiation exposure from clinical studies, including that from the present study, excluding background radiation but including diagnostic X-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. -

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Collier, MD, Principal Investigator — Quotient Clinical Ltd, Mere Way, Ruddington Fields, Nottingham, United Kingdom. NG11 6JS
Locations (1):
- Research Site, Nottingham, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 8 subjects were recruited into the study, as anticipated in the protocol. All received treatment with 20 mg [14C]-AZD9291 oral solution (free base equivalent) containing a nominal dose 1 μCi (0.037 MBq) activity as a single administration on Day 1 and all completed the study.
Pre-assignment Details: 8 evaluable patients were planned to be enrolled. These 8 evaluable patients were assigned to take 20 mg [14C]-AZD9291 oral solution (free base equivalent) containing a nominal dose 1 μCi (0.037 MBq) activity as a single administration on Day 1
Groups:
- AZD9291 20mg: 20 mg [14C]-AZD9291 oral solution (free base equivalent) containing a nominal dose 1 μCi (0.037 MBq) activity as a single administration on Day 1
Period: Overall Study
Arm/Group | AZD9291 20mg
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Radioactive Dose of [14C] Radiolabelled AZD9291 Recovered in Urine, Faeces, and in Total.
Description: The percentage of radioactive dose of [14C] radiolabelled AZD9291 recovered in urine, faeces, and in total, up to Day 85.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992. Urine (h): 0-4, 4-8, 8-12, 12-24, every 24 hrs to 504, 648-72, 816-40, 984-1008 and 1992-2016. Faeces: 0-24h and then as per urine.
Population: Pharmacokinetic population - all subjects who received 1 dose of [14C]-AZD9291 and had at least 1 postdose PK measurement without important protocol deviations/violations or events thought to significantly affect the PK of the investigational product
Measure: Mean (Standard Deviation); unit: Percentage radioactive dose recovered
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
Percentage radioactive dose recovered
  Urine | 14.2 (2.08)
  Faeces | 67.8 (4.35)
  Total | 81.9 (4.41)

2. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Area Under the Concentration-time Curve From Time Zero to the Time of the Last Quantifiable Concentration AUC(0-t)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of area under the concentration-time curve from time zero to the time of the last quantifiable concentration AUC(0-t), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
nM*h
  AZD9291 | 1580 (17.7) [799 to 2480]
  AZ5104 | 125 (17.4) [93.6 to 234]
  AZ7550 | 113 (15.6) [72.3 to 153]
  [14C] plasma | 178000 (15.2) [146000 to 227000]
  [14C] blood | 158000 (12.8) [135000 to 206000]

3. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Area Under the Concentration-time Curve From Time Zero to the Time of 72 Hours AUC(0-72)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of area under the concentration-time curve from time zero to the time of 72 hours AUC(0-72), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, 72
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
nM*h
  AZD9291 | 1010 (17.7) [632 to 1490]
  AZ5104 | 72.1 (17.4) [53.8 to 108]
  AZ7550 | 50.9 (15.6) [40.9 to 64.0]
  [14C] plasma | 9670 (15.2) [8060 to 12200]
  [14C] blood | 10700 (12.8) [8240 to 13200]

4. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Area Under the Concentration-time Curve From Time Zero to 24 Hours AUC(0-24)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of area under the concentration-time curve from time zero to the time of 24 hours AUC(0-24), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
nM*h
  AZD9291 | 444 (17.7) [318 to 632]
  AZ5104 | 24.4 (17.4) [17.3 to 36.6]
  AZ7550 | 15.7 (15.6) [12.1 to 20.5]
  [14C] plasma | 1980 (15.2) [1630 to 2420]
  [14C] blood | 2300 (12.8) [1840 to 2740]

5. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Maximum Plasma Concentration (Cmax)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of maximum plasma concentration (Cmax), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
nM
  AZD9291 | 29.9 (17.7) [22.3 to 38.5]
  AZ5104 | 1.41 (17.4) [.918 to 2.09]
  AZ7550 | .957 (15.6) [.804 to 1.34]
  [14C] plasma | 217 (15.2) [189 to 280]
  [14C] blood | 260 (12.8) [187 to 330]

6. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Time to Cmax (Tmax)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of by assessment of time to Cmax (tmax), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
hours
  AZD9291 | 6 (17.7) [6 to 8.12]
  AZ5104 | 6 (17.4) [6 to 36]
  AZ7550 | 36 (15.6) [6 to 48]
  [14C] plasma | 144 (15.2) [96 to 168]
  [14C] blood | 132.02 (12.8) [96 to 168.07]

7. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Lag Time Before Observation of Quantifiable Analyte Concentrations (Tlag)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of lag time before observation of quantifiable analyte concentrations (tlag), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
hours
  AZD9291 | 0 (17.7) [0 to 0]
  AZ5104 | .51 (17.4) [.5 to 1]
  AZ7550 | .76 (15.6) [0 to 1.5]
  [14C] plasma | 0 (15.2) [0 to 0]
  [14C] blood | .25 (12.8) [0 to .5]

8. Secondary Outcome: Pharmacokinetics of AZD9291 Plasma, Whole Blood and Plasma [14C] Radioactivity by Assessment of Apparent Oral Clearance (CL/F)
Description: Pharmacokinetics of AZD9291 plasma, whole blood and plasma [14C] radioactivity by assessment of apparent oral clearance (CL/F), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Mean (Full Range); unit: L/h
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
L/h
  AZD9291 | 26.7 (17.7) [16.1 to 49.9]
  [14C] plasma | .213 (15.2) [.165 to .262]
  [14C] blood | .231 (12.8) [.183 to .28]

9. Secondary Outcome: Pharmacokinetics of AZD9291 Plasma, Whole Blood and Plasma [14C] Radioactivity by Assessment of Apparent Volume of Distribution (Vz/F)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of apparent volume of distribution (Vz/F), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Mean (Full Range); unit: L
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
L
  AZD9291 | 2260 (17.7) [1630 to 3600]
  [14C] plasma | 146 (15.2) [117 to 168]
  [14C] blood | 191 (12.8) [128 to 230]

10. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Elimination Half-life (t1/2,λz)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of elimination half-life (t1/2,λz), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Mean (Full Range); unit: hour
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
hour
  AZD9291 | 61.2 (17.7) [48.2 to 77.5]
  AZ5104 | 55.2 (17.4) [41.3 to 77]
  AZ7550 | 82 (15.6) [60.2 to 100]
  [14C] plasma | 474 (15.2) [415 to 537]
  [14C] blood | 562 (12.8) [477 to 685]

11. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Elimination Rate Constant (λz)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of elimination rate constant (λz), derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 1/h
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
1/h
  AZD9291 | .0115 (17.7) [.00894 to .0144]
  AZ5104 | .0129 (17.4) [.00901 to .0168]
  AZ7550 | .00854 (15.6) [.00692 to .0115]
  [14C] plasma | .00147 (15.2) [.00129 to .00167]
  [14C] blood | .00125 (12.8) [.00101 to .00145]

12. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of AUC Metabolite to Parent Ratio, AZ7550 or AZ5104 AUC/AZD9291 AUC Adjusted for Differences in Molecular Weight (M/PAUC)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of AUC metabolite to parent ratio, AZ7550 or AZ5104 AUC/AZD9291 AUC adjusted for differences in molecular weight (M/PAUC), derived from the curves taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
Ratio
  AZ5104 | .0909 (17.4) [.0566 to .18]
  AZ7550 | .0848 (15.6) [.0635 to .162]

13. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Cmax Metabolite to Parent Ratio, AZ7550 or AZ5104 (M/PCmax)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of Cmax metabolite to parent ratio, AZ7550 or AZ5104 (M/PCmax), derived from the curves taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
ratio
  AZ5104 | .0471 (17.4) [.0346 to .0937]
  AZ7550 | .0319 (15.6) [.0232 to .0502]

14. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Cmax Ratio of Plasma AZD9291, AZ7550 or AZ5104 (PL) to Plasma Radioactivity (Cmax(PL)/Cmax(PR))
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of Cmax ratio of plasma AZD9291, AZ7550 or AZ5104 (PL) to plasma radioactivity (Cmax(PL)/Cmax(PR)), derived from the curves taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
ratio
  AZD9291 | .138 (17.7) [.117 to .199]
  AZ5104 | .00648 (17.4) [.00421 to .0109]
  AZ7550 | .0044 (15.6) [.00328 to .00586]

15. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Cmax Ratio of Whole Blood Radioactivity (WBR) to PR Cmax (WBR)/Cmax(PR)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of Cmax ratio of whole blood radioactivity (WBR) to PR Cmax (WBR)/Cmax(PR), derived from the curves taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
ratio | 1.2 (12.8) [.984 to 1.65]

16. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of AUC Ratio of Plasma AZD9291, AZD7550 or AZD5104 (PL) to Plasma Radioactivity (PR) AUC(PL)/AUC(PR)
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of AUC ratio of plasma AZD9291, AZD7550 or AZD5104 (PL) to plasma radioactivity (PR) AUC(PL)/AUC(PR), derived from the curves taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
ratio
  AZD9291 | .00826 (17.4) [.00429 to .0163]
  AZ5104 | .000751 (15.6) [.000508 to .00158]
  AZ7550 | .000698 (15.2) [.000566 to .00103]

17. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of AUC Ratio of WBR to PR (AUC(WBR)/AUC(PR))
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of AUC ratio of WBR to PR (AUC(WBR)/AUC(PR)), derived from the curves taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: ratio
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
ratio | .917 (12.8) [.809 to 1.06]

18. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Whole Blood and Plasma [14C] Radioactivity by Assessment of Area Under the Concentration-time Curve AUC
Description: Pharmacokinetics of AZD9291, its metabolites and whole blood and plasma [14C] radioactivity by assessment of area under the concentration-time curve AUC, derived from the curve taken during the treatment period.
Time Frame: Blood samples (hrs) - 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 18, 24, 36, 48, every 24 to 168, 336, 504, 648, 816, 904 and 1992.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM*h
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
nM*h
  AZD9291 | 1590 (17.7) [803 to 2490]
  AZ5104 | 143 (17.4) [106 to 242]
  AZ7550 | 132 (15.6) [92.5 to 170]
  [14C] plasma | 190000 (15.2) [153000 to 242000]
  [14C] blood | 174000 (12.8) [143000 to 219000]

19. Secondary Outcome: Pharmacokinetics of AZD9291, Its Metabolites and Urine [14C] Total Radioactivity by Assessment of Urine Concentration or Concentration Equivalent x Urine Volume (Aeu)
Description: Pharmacokinetics of AZD9291, its metabolites and urine [14C] total radioactivity by assessment of urine concentration or concentration equivalent x urine volume (Aeu), derived from the curve taken during the treatment period.
Time Frame: Urine (h): 0-4, 4-8, 8-12, 12-24, every 24 hrs to 504, 648-72, 816-40, 984-1008 and 1992-2016.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: nmol
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
nmol
  AZD9291 | 329 (133) [799 to 2480]
  AZ5104 | 167 (85.8) [93.6 to 234]
  AZ7550 | 184 (75.4) [72.3 to 153]
  [14C] urine | 3870 (673) [146000 to 227000]

20. Secondary Outcome: Pharmacokinetics of AZD9291 and Urine [14C] Total Radioactivity by Assessment of Percentage (or Fraction) of Actually Administered Dose / Radioactivity (Feu)
Description: Pharmacokinetics of AZD9291 and urine [14C] total radioactivity by assessment of percentage (or fraction) of actually administered dose / radioactivity (feu), derived from the curve taken during the treatment period.
Time Frame: Urine (h): 0-4, 4-8, 8-12, 12-24, every 24 hrs to 504, 648-72, 816-40, 984-1008 and 1992-2016.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of administered dose
Arm/Group | AZD9291 20mg
Number analyzed (Participants) | 8
Percentage of administered dose
  AZD9291 | .823 (.332) [799 to 2480]
  AZ5104 | .416 (.214) [93.6 to 234]
  AZ7550 | .460 (.189) [72.3 to 153]
  [14C] urine | 9.67 (1.69) [146000 to 227000]

ADVERSE EVENTS:
Time Frame: From screening through to day 85 (end of study)
Arm/Group | AZD9291 20mg
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 20mg (N=8)
Asthenopia (Eye disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Headache (Nervous system disorders) | 2 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hot flush (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent applications